CLINICAL TRIAL: NCT00780078
Title: Clinical Evaluation by Physical Therapist of Swallowing Disorders as a Predictor of Extubation Failure in Patients Intubated Orotracheally for Over 6 Days
Brief Title: Clinical Evaluation of Swallowing Disorders as a Predictor of Extubation Failure
Acronym: EVAKIN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: SCR060013; IRB00006477
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Central Nervous System Diseases; Acute Respiratory Failure; Shock; Heart Failure; Acute Poisoning
Keywords: Intensive care unit; Extubation failure; Physiotherapist; Pre-extubation bedside tests; Swallowing disorders
MeSH Terms: conditions — Central Nervous System Diseases; Shock; Heart Failure; Deglutition Disorders | interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients intubated orotracheally for over 6 days
  Interventions: Procedure: extubation

INTERVENTIONS:
Procedure: extubation — extubation failure in patients intubated orotracheally

SUMMARY:
Patients with failed extubation stay significantly longer in an intensive care unit (ICU) and have a higher mortality rate, than those intubated successfully. Reintubation is associated with life-threatening complications and a poor prognosis. Functional respiratory tests are frequently used as weaning parameters, however, they are not accurate enough to predict extubation failure. The incidence of swallowing dysfunction is underestimated, mainly among patients whose intubation lasts longer than 48 h.We previously observed that the assessment of the swallowing function and oropharyngeal motricity, conducted by the physiotherapist before extubation could be helpful for making decisions to extubate patients intubated for over 6 days. The objective of this study is to validate a scale previously devised and used for physiotherapist bedside evaluation of the swallowing function and oropharyngeal motricity, among patients intubated for over 6 days, to determine whether this scale is a good predictor of airway secretion-related extubation failure.Expected results : to validate a scale previously devised called " physiotherapist evaluation of the swallowing function and oropharyngeal motricity before extubation" by the mean of a multicentric study. In our hypothesis the clinical parameters studied could be predictive of extubation failure. Then, this evaluation could help the medical decision in the choice of the good time for extubation. The final objective is to lower the mortality related to extubation failure.

DETAILED DESCRIPTION:
* Patients selection, inclusion and procedure: All successive patients admitted to the medical or surgical ICU, and intubated by the orotracheal route for >6 days, will be prospectively enrolled when extubation will be decided. Patients with previous swallowing disorders, ENT surgery or chronic persistent vegetative status will not be included. All patients will have to fulfill the usual criteria for extubation. Then, before extubation, the different components of swallowing functions will be evaluated by the trained physiotherapist, using a bedside pre-extubation scale based on 3 tests: assessment of 1)- cervical, oral, labial and lingual motricity; 2)- the gag reflex; and 3)- swallowing. After extubation, the ability to cough and swallow, secretion volume, and the need for suctioning will be evaluated immediately, then at 24, 48 and 72 hours.
* Expected results : to validate a scale previously devised called " physiotherapist evaluation of the swallowing function and oropharyngeal motricity before extubation" by the mean of a multicentric study. In our hypothesis the clinical parameters studied could be predictive of extubation failure. Then, this evaluation could help the medical decision in the choice of the good time for extubation. The final objective is to lower the mortality related to extubation failure.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* patients intubated orotracheally for over 6 days
* patients fulfilling usual medical criteria for extubation, after a successful test of spontaneous ventilation, according to the French consensus conference (2001).

Exclusion Criteria:

* post ENT surgery- previous swallowing disorders
* chronic vegetative status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the objective of this study is to validate a scale previously devised and used for physiotherapist bedside evaluation of the swallowing function and oropharyngal motricity, among patients intubated for over 6 days, to determine whether this scale is a good predictor of airway secretion-related extubation failure
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Rate of reintubation within the 72 hours after extubation | 72 hours after extubation

SECONDARY OUTCOMES:
Delay for reintubation (hours) | 72 hours after extubation
Number of daily pharyngeal or tracheal suctioning | 72 hours after extubation
Pulmonary infection | 72 hours after extubation
Mortality | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Alain YELNIK, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE, Paris, France

REFERENCES:
- [Derived] Houze MH, Deye N, Mateo J, Megarbane B, Bizouard F, Baud FJ, Payen de la Garanderie D, Vicaut E, Yelnik AP; EVAKIN Study Group. Predictors of Extubation Failure Related to Aspiration and/or Excessive Upper Airway Secretions. Respir Care. 2020 Apr;65(4):475-481. doi: 10.4187/respcare.07025. Epub 2019 Nov 19. PMID 31744867